CLINICAL TRIAL: NCT05181787
Title: Biomarkers of Atrial Fibrillation Complicated With Stroke Based on Proteomics and Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yue LI (Other)
Responsible Party: Sponsor-Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: AF and stroke 1
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; Stroke; metabolomics; proteomics; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AF: Patients with AF
  Interventions: Diagnostic Test: Proteomics; Diagnostic Test: Metabolomics
- AF and stroke: Patients with AF complicated with stroke
  Interventions: Diagnostic Test: Proteomics; Diagnostic Test: Metabolomics

INTERVENTIONS:
Diagnostic Test: Proteomics — Proteomic data were obtained by LC-MS/MS Analysis-DIA platform.
Diagnostic Test: Metabolomics — Metabolomic data were obtained by UPLC-QTOF/MS platform.

SUMMARY:
Thrombus shedding in patients with atrial fibrillation (AF) can lead to cerebral artery embolism. Stroke caused by AF is very dangerous, which not only threatens the life of patients, but also seriously affects the quality of life. This study aims to explore the biomarkers of stroke in patients with AF by integrating proteomics and metabolomics data, and establish the network relationship of stroke in patients with AF, so as to reveal the molecular mechanism of stroke in patients with AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Admission with atrial fibrillation or clinic visit for atrial fibrillation
3. Receive routine anticoagulant therapy;
4. Signing the consent form

Exclusion Criteria:

1. Pregnant women;
2. Lactating women;
3. Severe mitral stenosis;
4. Severe impairment of liver function;
5. Severe renal insufficiency;
6. Thyroid dysfunction requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The blood samples of patients with AF and patients with AF complicated with stroke were taken. The supernatant was centrifuged and put into - 80 ℃ refrigerator for storage.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of atrial fibrillation complicated with stroke based on proteomics and metabolomics | 1 day
  By combining proteomics and metabolomics data, the investigators were able to identify the common pathways involved in AF with stroke.

SECONDARY OUTCOMES:
Quantitative changes of individual metabolites and proteins were calculated and graphed using the KEGG mapping tools. | 1 day
By combining proteomics and metabolomics data, the investigators were able to identify the common pathways involved in AF with stroke. | 1 day
All of the omics data were used to compare proteins/enzymes with metabolic pathways. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Yan, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided